CLINICAL TRIAL: NCT01915992
Title: Natural Killer Cells Functions, Tumoral Escape to Immune System and Regulation of Natural Cytotoxixity Receptors in Haematological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012-A01412-41; 2012-34 (Other: AP HM)
Record Dates: First submitted 2013-02-20; First posted 2013-08-05 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volunteer healthy (Other)
  Interventions: Other: blood samples
- leukemia patient's (Active Comparator)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples

SUMMARY:
The NK cells participate in the innate immunity against infectious agents or transformed cells that are recognized as "no self" by the absent, weak or abnormal expression of human leukocyte antigen (HLA) class I molecules. According to the "missing self hypothesis", a negative signal is delivered to NK cells when their inhibitory receptors are engaged by the specific HLA class I molecules. NK activation requires a positive signal delivered by the engagement of activating receptors, more particularly of the "Natural cytotoxicity receptors" or NCRs who are directly involved in the natural cytotoxicity of Natural Killer. The activating receptors include NKp46, NKp44 and NKp30, also called NCR 1, 2 and 3 respectively. NKp46 and NKp30 are constitutively expressed on the surface of the NK, the expression of NKp44 is observed only after activation of cells NK. NK cells from most (80%) healthy donors express a high quantity of NCR on their surface, corresponding to the NCRbright phenotype while only 20 % present the NCRdull phenotype. In sharp contrast, most patients (80%) having leukaemia have the NCRdull while only 20 % patients have the NCRbright phenotype. The culture of NK from healthy donors ( NCRbright) with leukaemic cells result in decreased expression of the NKp30 while there is no difference on expression if these same NK are cultivated with cells from healthy donors. Moreover, study of AML patients showed that the NCRdull phenotype was acquired during leukemia development because it was observed its complete (for NKp46) or partial (for NKp30) reversibility in patients achieving complete remission (CR). Reversibility of the NCRdull phenotype after CR suggested that leukemia cells might be involved in NCR down-regulation. In line with these observations, we aim to study the mechanism of NCR down-regulation by cultivating NK NCRbright from healthy donors with leukaemic cells or healthy haematopoietic cells, in order to observe the appearance of the NCRdull phenotype and verify by qPCR if this down-regulation is transcriptionnal. If this hypothesis is be verified, we will study the regulation of NCR by focusing on the implication of genes NCR transcription factors via bio-informatic analysis of putative transcription factors fixation sequences in the promoters of these genes, followed by the verification of the capacity of identified sequences to bind transcription factors. Ultimately, we will verify the real implications of these transcription factors by studying the effect of their silencing by RNA interference experiments.

ELIGIBILITY:
Inclusion Criteria:

* Grown-up patients having a leukaemia aigue myéloïde (LAM) in the diagnosis, whatever is LAM's subcategory (FAB or cytogenetics).
* The patients that must be informed at the same time, willing, and having given their agreement in writing.

Exclusion Criteria:

* Refusal of the patient.
* Phénotypage NK not corresponding to the quotas dull / bright required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-08 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
blood sample | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France